CLINICAL TRIAL: NCT00685802
Title: A Comparative Bioavailability Study of Cilostazol Tablets, 50mg, Under Fasting Conditions
Brief Title: Fasted Bioavailability Study of Cilostazol Tablets, 50mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 11801
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2009-12-22 (Estimated); Status verified 2009-11

CONDITIONS: Therapeutic Equivalency, Healthy
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol 50 mg Tablets (Experimental): A single dose of cilostazol (2 x 50 mg tablets) administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Cilostazol 50 mg Tablets
- Cilostazol (Pletal® ) 50 mg Tablets (Experimental): A single dose of Cilostazol (Pletal® tablets, 2 x 50 mg ) administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Cilostazol (Pletal®) 50 mg Tablets

INTERVENTIONS:
Drug: Cilostazol 50 mg Tablets — Cilostazol (2 x 50 mg tablets) administered after an overnight fast of at least 10 hours
  Arms: Cilostazol 50 mg Tablets
Drug: Cilostazol (Pletal®) 50 mg Tablets — Cilostazol (Pletal® Tablets, 2 x 50mg) administered after an overnight fast of at least 10 hours.
  Other Names: Pletal®
  Arms: Cilostazol (Pletal® ) 50 mg Tablets

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of a test formulation of cilostazol tablets to an equivalent dose of Pletal® (cilostazol) tablets after a single oral dose administered under fasting conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of a test formulation of cilostazol tablets to an equivalent dose of Pletal® (cilostazol) tablets after a single oral dose administered under fasting conditions. Thirty-two non-smoking, non-obese, healthy male and female volunteers between the ages of 18 and 55 will be randomly assigned in a crossover fashion to receive each of two cilostazol dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive either a single oral dose of the test formulation, cilostazol (2 x 50 mg tablets), or a single oral dose of the reference formulation, Pletal® (2 x 50 mg tablets). After a 7 day washout period on the morning of Day 8, following an overnight fast of at least 10 hours, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of cilostazol. Blood sampling will then continue on a non-confined basis at 36 and 48 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Blood pressure and pulse will be measured before dosing and at 3 and 24 hours post-dose. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-55 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* No more than 15% plus or minus from ideal weight for subject's height and elbow breadth as defined by the Metropolitan Life Insurance Company Statistical Bulletin. Extrapolations, if required, to be conducted according to BASi Standard Operating Procedures
* Medically healthy on the basis of medical history and physical examination within 30 days prior to the start of the study
* Test results from blood chemistry, hematology, and urinalysis performed within 30days prior to the start of the study within clinically acceptable limits
* At screening, subjects must have blood pressure and pulse rate within the following ranges: Systolic blood pressure 90-140mmHg; Diastolic blood pressure 50-90mmHg; Pulse 45-100 bpm
* An acceptable electrocardiogram (EKG): sinus rhythm with no evidence of AV block or ischemic changes

Exclusion Criteria:

* Prescription drug use (excluding hormonal contraceptives) within 14 days prior to drug administration, each period
* Aspirin ingestion within 7 days prior to drug administration, each period
* Use of any over-the-counter preparations, herbal remedies, and/or nutritional supplements within 7 days prior to drug administration, each period
* Consumption of grapefruit juice or grapefruit-containing products within 72 hours prior to drug administration , each period
* Consumption of alcohol within 24 hours prior to drug administration, each period
* Consumption of caffeine within 10 hours prior to drug administration, each period
* Female subjects must not be pregnant or nursing; and must be surgically sterile; one year post-menopausal; or on hormonal contraceptive agent(s), a diaphragm or condom with spermicidal foam or jelly, or IUD for at least three months prior to drug administration and agree to use the same method of contraception for at least 1 month after the last drug administration
* Subjects with a history or presence of significant organ system (cardiovascular, neurological, hepatic, hematopoietic, renal, pulmonary, endocrine, or gastrointestinal) disorders, or ongoing infectious diseases
* History of hypersensitivity or adverse reactions to cilostazol (Pletal®), or other related drugs
* Recent (12 month) history or evidence of alcoholism or drug abuse
* Positive urine screening of drugs of abuse
* Positive results to Human Immunodeficiency Virus (HIV) or Hepatitis B surface Antigen (HBsAg) tests
* Participation in another clinical trial in the previous 30 days before day 1 of this study
* Donation of blood in the previous 30 days before day 1 of this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-06; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilip K Guha-Ray, M.D., Principal Investigator — BASi Baltimore Clinical Research Unit

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-two healthy adult male and female volunteers from the community-at-large were enrolled.
Groups:
- Cilostazol 50 mg Tablets Then Pletal® 50 mg Tablets: On the morning of Day 1 subjects received two tablets of the test formulation, Cilostazol 50 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received two tablets of the reference formulation, Pletal® 50 mg, after an overnight fast of at least 10 hours.
- Pletal® 50 mg Tablets Then Cilostazol 50 mg Tablets: On the morning of Day 1 subjects received two tablets of the reference formulation, Pletal® 50 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received two tablets of the test formulation, Cilostazol 50 mg, after an overnight fast of at least 10 hours.
Period: First Intervention
Arm/Group | Cilostazol 50 mg Tablets Then Pletal® 50 mg Tablets | Pletal® 50 mg Tablets Then Cilostazol 50 mg Tablets
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Cilostazol 50 mg Tablets Then Pletal® 50 mg Tablets | Pletal® 50 mg Tablets Then Cilostazol 50 mg Tablets
Started | 16 | 16
Completed | 14 | 15
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Cilostazol 50 mg Tablets Then Pletal® 50 mg Tablets | Pletal® 50 mg Tablets Then Cilostazol 50 mg Tablets
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cilostazol 50 mg Tablets and Pletal® 50 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received two tablets of either Cilostazol 50 mg or Pletal® 50 mg following an overnight fast of at least 10 hours.
Arm/Group | Cilostazol 50 mg Tablets and Pletal® 50 mg Tablets
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.25 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that cilostazol (test and reference product) reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 16, 24, 36 and 48 hours after drug administration.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cilostazol 50 mg Tablets; Pletal® 50 mg Tablets: On the morning of Day 1 subjects received two tablets of either the test formulation, cilostazol 50mg, or the reference formulation, Pletal® 50 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received the alternate regimen following an overnight fast of at least 10 hours.
Arm/Group | Cilostazol 50 mg Tablets | Pletal® 50 mg Tablets
Number analyzed (Participants) | 29 | 29
ng/mL | 565.52 (155.67) | 570.60 (174.72)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Cilostazol 50 mg Tablets | Pletal® 50 mg Tablets
Number analyzed (Participants) | 29 | 29
ng-hr/mL | 7,265.38 (1,975.87) | 7,354.03 (2,048.83)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses of cilostazol and Pletal® are based on 28 and 27 subjects, respectively. Reliable estimates could not be obtained for one subject administered Cilostazol and two subjects administered Pletal® because there was not a smooth decline in concentrations in the terminal phase of elimination.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Cilostazol 50 mg Tablets | Pletal® 50 mg Tablets
Number analyzed (Participants) | 28 | 27
ng-hr/mL | 8,641.26 (3,010.04) | 8,706.54 (3,142.36)

ADVERSE EVENTS:
Time Frame: All adverse events were recorded during the 14 day course of the study.
Groups:
- Cilostazol 50 mg Tablets; Pletal® 50 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received two tablets of either cilostazol 50 mg or Pletal® 50 mg following an overnight fast of at least 10 hours.
Arm/Group | Cilostazol 50 mg Tablets | Pletal® 50 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 10/31 | 12/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3.22% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol 50 mg Tablets (N=31) | Pletal® 50 mg Tablets (N=30)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — decreased pulse-heart rate
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) — elevated systolic
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) — elevated pulse
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — decreased hematocrit
Anemia hypochrom (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — decreased hemoglobin
hypotension (Cardiac disorders) | 1 (1) | 0 (0) — low diastolic
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — increased absolute neutrophils, increased white blood cell count
Albuminuria (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — protein 1+ urine
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — elevated glucose
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — pain in left wrist
paresthesia circumoral (Nervous system disorders) | 1 (1) | 0 (0) — abnormal sensation of lips
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — sore throat
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — congestion, post-nasal drip
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) — urine blood 3+
Urine abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) — leukocyte 2+

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days